CLINICAL TRIAL: NCT04958421
Title: A Randomized, Controlled, Pilot Study to Evaluate Safety and Feasibility of Pressure-controlled Intermittent Coronary Sinus Occlusion (PiCSO) Therapy in Patients With ST Elevation Inferior Wall Myocardial Infarction Presenting With TIMI 0 or 1 and Symptom Duration ≤ 12 Hours Treated Adjunct to Percutaneous Coronary Intervention (PCI) Compared to Standard PCI.
Brief Title: A Study to Evaluate Safety and Feasibility of PiCSO Therapy in Patients With ST Elevation Inferior Wall Myocardial Infarction.
Acronym: PiCSO-AMI-V
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated due to lack of financing
Sponsor: Miracor Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIR-CIP 0005
Record Dates: First submitted 2021-06-29; First posted 2021-07-12 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2022-04

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Inferior Wall Myocardial Infarction
Keywords: PiCSO; PiCSO Impulse System
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Inferior Wall Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: Prospective, multicenter, randomized, controlled, parallel-groups, pilot stage study
Who Masked: Outcomes Assessor
Masking Description: Analysis of the secondary efficacy endpoint, changes in left and right ventricular function, will be analyzed by an independent Corelab, blinded to the allocated treatment arm.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This is the actual control group receiving conventional therapy, ie. percutaneous coronary intervention.
- PiCSO (Experimental): This arm will be treated with Pressure controlled intermittent Coronary Sinus Occlusion (PiCSO) in addition to conventional therapy (percutaneous coronary intervention).
  Interventions: Device: PiCSO Impulse System

INTERVENTIONS:
Device: PiCSO Impulse System — After blood flow restoration, the subjects meeting all eligibility criteria will be enrolled into the study and randomized either to PiCSO Group or Control Group. If the subject is randomized to PiCSO Group, the coronary sinus (CS) will be cannulated through the femoral vein and the PiCSO Impulse Catheter will be placed in the CS. Once PiCSO Impulse Catheter is placed into CS, PiCSO treatment is started followed by stenting. The physician shall target a PiCSO treatment of 45 minutes whereas the treatment should be continued during and post stent insertion. At the end of the PiCSO treatment, the PiCSO Impulse Console is stopped and the PiCSO Impulse Catheter is removed.
  Arms: PiCSO

SUMMARY:
The objective of this study is to assess safety and feasibility of Pressure-controlled intermittent Coronary Sinus Occlusion (PiCSO) therapy in patients with extensive ST elevation inferior wall myocardial infarction presenting with TIMI 0 or 1 and symptom duration ≤ 12 hours undergoing percutaneous coronary intervention (PCI) compared to standard PCI.

DETAILED DESCRIPTION:
This is a multicenter, randomized (2 PiCSO :1 Control), controlled, pilot study to evaluate safety and feasibility of Pressure-controlled intermittent Coronary Sinus Occlusion (PiCSO) therapy in patients with extensive ST elevation inferior wall myocardial infarction presenting with TIMI 0 or 1 and symptom duration ≤ 12 hours treated adjunct to percutaneous coronary intervention (PCI) compared to standard PCI. Patients with an ST-segment elevated inferior infarct eligible for PCI will be invited to participate in the PiCSO-AMI-V Inferior STEMI study. After consent as per approved ethics committee requirements, baseline assessments will be performed. PCI of the culprit vessel should be performed per standard practices. After TIMI flow restoration, the subjects meeting all eligibility criteria will be enrolled into the study and randomized either to PiCSO Group or Control Group. If the subject is randomized to PiCSO Group, the coronary sinus (CS) will be cannulated through the femoral vein and the PiCSO Impulse Catheter will be placed in the CS. In the event the PiCSO Impulse Catheter cannot be placed in the CS within 30 minutes, the physician should proceed with the regular PCI and the PiCSO treatment will be considered a failure. Once PiCSO Impulse Catheter is placed into CS, PiCSO treatment is started followed by stenting. The physician shall target a PiCSO treatment of 45 minutes whereas the treatment should be continued during and post stent insertion. At the end of the PiCSO treatment, the PiCSO Impulse Console is stopped and the PiCSO Impulse Catheter is removed. The patient is seen for a FU visit at 12-36 hours, 30 days, 6 months and 1 year post index procedure. 12-36 hours and 6 months post index the patient will get a echocardiogram. At every FU visit safety data and health status will be documented.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Right dominance with culprit lesion in mid or proximal RCA
3. Pre-PCI TIMI flow 0 or 1 in the culprit lesion
4. Symptom onset time consistent with myocardial ischemia (e.g. persistent chest pain, shortness of breath, nausea/vomiting, fatigue, palpitations or syncope) ≤ 12 h
5. ECG evidence of acute inferior myocardial infarction with ST-elevation ≥ 2 mm (0.2 mV) in 2 or more contiguous inferior precordial ECG leads (II, III, AVF) in men or ≥ 1.5 mm (0.15 mV) in women
6. Emergent PCI will be performed according to national and local hospital guidelines
7. Consent per approved national EC specific requirements prior to the procedure.

Exclusion Criteria:

1. Patient transferred from an outside hospital where invasive coronary procedure was attempted (including diagnostic catheterization)
2. Implants or foreign bodies in the coronary sinus
3. Left main disease >= 50%
4. Large left anterior descending artery providing blood supply beyond the left ventricular apex (supplying part of the inferior wall) as judged by angiography.
5. Known allergy to polyurethanes, PET or stainless steel, both heparin and bivalirudin, or all of clopidogrel, ticagrelor or prasugrel that cannot be adequately premedicated
6. Known pregnancy or breastfeeding
7. Known large pericardial effusion or cardiac tamponade
8. Known hemodynamically relevant left to right and right to left shunt
9. Previous CABG
10. Known neurologic abnormality such as tumor or AV malformation, history of stroke within 6 months, any prior intracranial bleed or any permanent neurologic defect
11. History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), any recent GU or GI bleed (within 3 months)
12. Administration of fibrinolytic therapy within 24 hours prior to enrollment
13. Cardiogenic shock (SBP < 90 mmHg), need for mechanical circulatory support, intravenous pressor or pre-randomization intubation
14. Patients with cardio-pulmonary resuscitated (CPR) cardiac arrest for more than 5 min or whom baseline neurologic status is not present
15. Patient not suitable for femoral vein access
16. Active participation in another drug or device investigational study that has not reached its primary endpoint
17. Known severe kidney disease (eGFR <=30 mL/min/1.73 m2 by MDRD formula) or on hemodialysis
18. COPD with home oxygen therapy or on chronic steroid therapy for COPD
19. Unconscious on presentation
20. Patients under judicial protection, legal guardianship or curatorship
21. Patient has other medical illness (e.g., cancer, dementia) or known history of substance abuse (alcohol, cocaine, heroin, etc.) that may cause non-compliance with the protocol, confound the data interpretation, or is associated with limited life expectancy of less than 1 year
22. Patients with definite or probable COVID-19 diagnosis > 4 weeks prior to the current MI unless they had returned to their baseline state of health after recovery from the COVID-19 illness
23. Any evidence of active infectious disease, or definite or probable COVID-19 diagnosis within the prior 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Adverse Device Effect (ADE) rate at 30 days post index procedure | 30 days post MI
  Adverse Device Effect (ADE) rate at 30 days post index procedure

SECONDARY OUTCOMES:
A severity index derived as the mean wall motion score within the region of AWM | 12 to 36 hours and 6 months post MI
  1. Changes in left and right ventricular function assed by echocardiogram performed within 12 to 36 hours of index PCI and 6 months post index PCI
Ejection fraction using measured by Simpson's method with 2 apical view | 12 to 36 hours and 6 months post MI
  1. Changes in left and right ventricular function assed by echocardiogram performed within 12 to 36 hours of index PCI and 6 months post index PCI
The absolute size of the region of abnormal wall motion (AWM) | 12 to 36 hours and 6 months post MI
  1. Changes in left and right ventricular function assed by echocardiogram performed within 12 to 36 hours of index PCI and 6 months post index PCI
Percentage of the endocardium involved (%AWM) | 12 to 36 hours and 6 months post MI
  1. Changes in left and right ventricular function assed by echocardiogram performed within 12 to 36 hours of index PCI and 6 months post index PCI
Wall motion score | 12 to 36 hours and 6 months post MI
  1. Changes in left and right ventricular function assed by echocardiogram performed within 12 to 36 hours of index PCI and 6 months post index PCI
hs-Troponin | hospital admission, 6h, 12h, 24h and then daily until day 5 after PCI or discharge
  Maximum and AUC of hs-Troponin
C-reactive protein | hospital admission, 6h, 12h, 24h and then daily until day 5 after PCI or discharge
  Maximum, AUC and velocity of C-reactive protein
CK-MB | hospital admission, 6h, 12h, 24h and then daily until day 5 after PCI or discharge
  Maximum and AUC of CK-MB
Blushing index | Immediately after treatment
  Blushing index at the end of the procedure
ST-segment resolution | 60-90 minutes post flow restoration
  ST-segment resolution at 60-90 minutes post flow restoration
Device success and procedural success rate presented as % of subjects | 1 day
  Device and Procedural success, assessed as percent of subjects with successful access, delivery, and retrieval of the device and its delivery system

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Banning, Prof., Principal Investigator — John Radcliffe Hospital, Oxford
Locations (11):
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus
  - Odense Universitetshospital, Odense
- France (3):
  - CHU Hôpiteaux de Bordeaux, Hôpital Haut Lévéque, Bordeaux
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Switzerland (2):
  - Bern University Hospital, Bern
  - EOC Ospedale Regionale di Lugano - Civico, Lugano
- United Kingdom (3):
  - Golden Jubilee National Hospital, Clydebank
  - New Edinburgh Royal Infirmary, Edinburgh
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No